CLINICAL TRIAL: NCT01794507
Title: A Phase 1b Study Evaluating the Safety and Pharmacokinetics of ABT-199 in Relapsed or Refractory Multiple Myeloma Subjects Who Are Receiving Bortezomib and Dexamethasone as Their Standard Therapy
Brief Title: A Study Evaluating ABT-199 in Multiple Myeloma Subjects Who Are Receiving Bortezomib and Dexamethasone as Standard Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-901; 2011-004626-10 (EudraCT Number)
Record Dates: First submitted 2012-12-13; First posted 2013-02-20 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: relapsed/refractory multiple myeloma; relapsed multiple myeloma; refractory multiple myeloma; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — venetoclax; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABT-199 + BTZ/Dex Dose Escalation Cohorts (Experimental): Evaluate the safety and pharmacokinetics profile of ABT-199 administered with standard therapy bortezomib and dexamethasone in a dose escalation scheme in approximately 54 subjects.
  Interventions: Drug: ABT-199; Drug: bortezomib; Drug: dexamethasone
- ABT-199 + BTZ/Dex Safety Expansion Cohort (Experimental): Safety expansion cohort to further evaluate recommended phase two dose (RPTD) of ABT-199 administered with standard therapy bortezomib and dexamethasone in approximately 12 subjects.
  Interventions: Drug: ABT-199; Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: ABT-199 — ABT-199 at cohort-defined dosing schedules and dose levels. ABT-199 at defined dose and schedule for Safety Expansion cohort
Drug: bortezomib — Bortezomib at cohort-defined dosing schedules and dose levels. Bortezomib at defined dose and schedule for Safety Expansion cohort
Drug: dexamethasone — Dexamethasone at cohort-defined dosing schedules and dose levels. Dexamethasone at defined dose and schedule for Safety Expansion cohort.

SUMMARY:
The primary objectives of this study are to assess the safety profile, characterize pharmacokinetics (PK) and determine the dosing schedule, maximum tolerated dose (MTD), and the recommended phase two dose (RPTD) of ABT-199 when administered in subjects with relapsed /refactory multiple myeloma who are receiving bortezomib and dexamethasone as their standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance score less than or equal to 1
* Diagnosis of multiple myeloma previously treated with at least 1 prior line of therapy (dose escalation only) or (safety expansion only) received treatment with a proteasome inhibitor or an IMiD(r) or immunomodulatory agent (e.g., thalidomide, lenalidomide). Induction therapy and following stem cell transplant are considered a single line of therapy.
* Measurable disease at Screening: Serum monoclonal protein greater than or equal to 1 g/dL by protein electrophoresis, or greater than or equal to 200 mg monoclonal protein in the urine on 24-hr electrophoresis, or serum immunoglobulin free light chain greater than or equal to 10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio.
* Subjects with a history of autologous or allogenic stem cell transplant must have adequate bone marrow independent of any growth factor support, and have recovered from any transplant related toxicity(s); and either greater than 100 days post-autologous transplant (prior to first dose of study drug) or greater than or equal to 6 months post-allogenic transplant (prior to first dose of study drug) and not have active graft-versus-host disease (i.e., requiring treatment).
* Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening.

Exclusion Criteria:

* Exhibits evidence of other clinically significant uncontrolled condition(s), including, but not limited to: uncontrolled systemic infection (viral, bacterial, or fungal), diagnosis of fever and neutropenia within 1 week prior to first dose of study drug
* Cardiovascular disability status of New York Heart Association Class greater than or equal to 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea or anginal pain.
* Significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, pulmonary or hepatic disease, that in the opinion of the investigator, would adversely affect his/her participation in the study.
* History of other active malignancies other than multiple myeloma within the past 3 years prior to study entry, with the following exceptions: adequately treated in situ carcinoma of the cervix uteri, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin, previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Tested positive for HIV or hepatitis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-11-19 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Determination of peak concentration (Cmax) of ABT-199 | Approximately 5 days in Cycle 1 then on Day 1 of Cycles 2,4,6,8
  Blood samples for pharmacokinetic analysis of ABT-199 will be collected at designated timepoints
Determine maximum tolerated dose (MTD), and recommended phase two dose (RPTD) of ABT-199 | Minimum first cycle of dosing (21 days)
  ABT-199 will be dose-escalated until the largest dose is reached that is determined to be safe based on adverse event reporting and dose-limiting toxicities information from all subjects.
Number of participants with adverse events | From subject's first dose of ABT-199 until 30 days after subject's last dose of ABT-199; up to 2 years following last subject first dose.
  Collect all adverse events at each visit.
Determination of trough concentration (Ctrough) of ABT-199 | Approximately 5 days in Cycle 1 then on Day 1 of Cycles 2,4,6,8
  Blood samples for pharmacokinetic analysis of ABT-199 will be collected at designated timepoints
Determination of area under the concentration versus time curve (AUC) of ABT-199 | Approximately 5 days in Cycle 1 then on Day 1 of Cycles 2,4,6,8
  Blood samples for pharmacokinetic analysis of ABT-199 will be collected at designated timepoints
Determine recommended phase two dose (RPTD) of ABT-199 | Minimum first cycle of dosing (21 days
  ABT-199 will be dose-escalated until the largest dose is reached that is determined to be safe based on adverse event reporting and dose-limiting toxicities information from all subjects.

SECONDARY OUTCOMES:
Duration of Response | Measured up to 48 months after the last subject has enrolled in the study
  Number of days from the day of initial response is objectively documented to the day that disease progression is objectively documented
Objective Response Rate | Measured up to 48 months after the last subject has enrolled in the study
  The proportion of subjects with response using International Myeloma Working Group (IMWG) response criteria will be computed for all subjects with active disease at baseline (in the opinion of the investigator)
Time to Disease Progression | Measured up to 48 months after the last subject has enrolled in the study
  Number of days from the date of the first dose of ABT-199 to the date of the subject's disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (9):
- United States (5):
  - University of Arizona Cancer Center - North Campus /ID# 117876, Tucson, Arizona
  - Mayo Clinic /ID# 121495, Jacksonville, Florida
  - Northwestern University Feinberg School of Medicine /ID# 117477, Chicago, Illinois
  - University of Michigan Hospitals /ID# 80353, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 77235, Rochester, Minnesota
- Australia (2):
  - Peter MacCallum Cancer Ctr /ID# 79553, Melbourne, Victoria
  - Royal Melbourne Hospital /ID# 79533, Parkville, Victoria
- France (2):
  - CHRU Lille - Hôpital Claude Huriez /ID# 77234, Lille, Hauts-de-France
  - CHU de Nantes, Hotel Dieu -HME /ID# 78773, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau P, Chanan-Khan A, Roberts AW, Agarwal AB, Facon T, Kumar S, Touzeau C, Punnoose EA, Cordero J, Munasinghe W, Jia J, Salem AH, Freise KJ, Leverson JD, Enschede SH, Ross JA, Maciag PC, Verdugo M, Harrison SJ. Promising efficacy and acceptable safety of venetoclax plus bortezomib and dexamethasone in relapsed/refractory MM. Blood. 2017 Nov 30;130(22):2392-2400. doi: 10.1182/blood-2017-06-788323. Epub 2017 Aug 28. PMID 28847998
- [Derived] Matulis SM, Gupta VA, Nooka AK, Hollen HV, Kaufman JL, Lonial S, Boise LH. Dexamethasone treatment promotes Bcl-2 dependence in multiple myeloma resulting in sensitivity to venetoclax. Leukemia. 2016 May;30(5):1086-93. doi: 10.1038/leu.2015.350. Epub 2015 Dec 28. PMID 26707935